CLINICAL TRIAL: NCT05147129
Title: Characterizing the Microbiome in Postmenopausal Women With Vulvar Lichen Sclerosus
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Dermatology Foundation (Other)
Responsible Party: Principal Investigator, Melissa Mauskar, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU2021-0392
Record Dates: First submitted 2021-10-26; First posted 2021-12-07 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Vulvar Lichen Sclerosus
MeSH Terms: conditions — Vulvar Lichen Sclerosus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postmenopausal with vulvar lichen sclerosus: Includes postmenopausal patients with clinically-active vulvar lichen sclerosus, as determined by biopsy or examination by a vulvar specialist
- Postmenopausal without vulvar lichen sclerosus: Includes postmenopausal patients without vulvar lichen sclerosus

SUMMARY:
Vulvar lichen sclerosus (LS) is a chronic inflammatory disease, often diagnosed at late stages after scarring has obliterated normal vulvar architecture and severely affected a woman's quality of life. First line therapy for vulvar LS is ultrapotent topical steroids. If left untreated, this condition can cause complete stenosis of the vaginal introitus and 5% of patients may develop squamous cell carcinoma (SCC).

Lichen sclerosus is more common in pre-pubertal children and in post-menopausal women suggesting that hormonal shifts may contribute to disease pathogenesis. Small studies in children with LS have also shown that the microbiome is altered in LS. Little is known about the skin microbiota in postmenopausal patients with vulvar LS.

To determine if the microbiome is altered in vulvar skin of postmenopausal patients with LS, this study will use 16s sequencing to broadly characterize the microbiota of vulvar skin with LS compared to control vulvar skin. The study team hypothesizes that patients with vulvar LS will have a unique vulvar microbial signature compared to age-matched controls. This study also seeks to elucidate differences in the vulvar microbiome of patients with LS after treatment of their underlying condition. The study team hypothesizes that the vulvar microbiome will change after treatment for vulvar LS.

Vulvar dermatoses are an understudied area in dermatology with limited therapeutic options. Innumerable women often suffer in silence with vulvar LS. The long-term goal of this work is to understand factors that contribute to vulvar LS so that intervention may be undertaken before irreversible scarring and SCC develop.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal

Exclusion Criteria:

* Use of systemic hormone replacement
* Use of antibiotics in prior three months
* Urinary incontinence, which is defined by: 1) two incontinence episodes in the past three days and also 2) regular incontinence over the past three months that has necessitated use of incontinence protection garments

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Group - Postmenopausal with vulvar lichen sclerosus: selected from patients presenting to vulvar dermatology clinic
  Group - Postmenopausal without vulvar lichen sclerosus: selected from dermatology or gynecology clinics
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Operational taxonomic unit (OTU) relative abundance | Baseline
  Similar 16s sequencing reads will be clustered into OTUs and relative abundance of OTUs in the samples under investigation will be reported
Operational taxonomic unit (OTU) relative abundance | 10-14 weeks after beginning treatment for vulvar lichen sclerosus, if applicable
  Similar 16s sequencing reads will be clustered into OTUs and relative abundance of OTUs in the samples under investigation will be reported

SECONDARY OUTCOMES:
Alpha and beta diversity | Baseline
  Alpha and beta diversity will be estimated in the context of sample metadata
Alpha and beta diversity | 10-14 weeks after beginning treatment for vulvar lichen sclerosus, if applicable
  Alpha and beta diversity will be estimated in the context of sample metadata

CONTACTS AND LOCATIONS:
Overall Officials: Melissa M Mauskar, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee A, Bradford J, Fischer G. Long-term Management of Adult Vulvar Lichen Sclerosus: A Prospective Cohort Study of 507 Women. JAMA Dermatol. 2015 Oct;151(10):1061-7. doi: 10.1001/jamadermatol.2015.0643. PMID 26070005
- [Background] Melnick LE, Steuer AB, Bieber AK, Wong PW, Pomeranz MK. Lichen sclerosus among women in the United States. Int J Womens Dermatol. 2020 May 8;6(4):260-262. doi: 10.1016/j.ijwd.2020.05.001. eCollection 2020 Sep. PMID 33015282
- [Background] Mauskar MM, Marathe K, Venkatesan A, Schlosser BJ, Edwards L. Vulvar diseases: Conditions in adults and children. J Am Acad Dermatol. 2020 Jun;82(6):1287-1298. doi: 10.1016/j.jaad.2019.10.077. Epub 2019 Nov 8. PMID 31712170
- [Background] Chattopadhyay S, Arnold JD, Malayil L, Hittle L, Mongodin EF, Marathe KS, Gomez-Lobo V, Sapkota AR. Potential role of the skin and gut microbiota in premenarchal vulvar lichen sclerosus: A pilot case-control study. PLoS One. 2021 Jan 14;16(1):e0245243. doi: 10.1371/journal.pone.0245243. eCollection 2021. PMID 33444404